CLINICAL TRIAL: NCT02131493
Title: A Open-label, Randomized Study of S-1 and and Gemcitabine vs Gemcitabine Alone as Adjuvant Therapy for Patients With Resected Pancreatic Cancer
Brief Title: S-1 and and Gemcitabine vs Gemcitabine Alone as Adjuvant Chemotherapy for Patients With Resected Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, First affiliated hospital, Zhejiang university, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYYYMedOncoPAC01
Record Dates: First submitted 2014-05-03; First posted 2014-05-06 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination); Gemcitabine

ARMS (2):
- Gemcitabine (Active Comparator): Gemcitabine：1000mg/m2，iv 30min，d1, d8,d15 q4w, 6 cycles
  Interventions: Drug: S-1, Gemcitabine
- S-1+ Gemcitabine (Experimental): S-1：40~60mg bid，d1~14; (S-1 dosage：BSA <1.25m2，40mg bid，1.25m2≤BSA≤1.5m2，50mg bid，BSA>1.5m2， 60mg bid) Gemcitabine：1000mg/m2，iv 30min，d1, d8 q3w, 8 cycles
  Interventions: Drug: S-1, Gemcitabine

INTERVENTIONS:
Drug: S-1, Gemcitabine

SUMMARY:
This study is a randomized, open-label, controlled study that will compare the efficacy of S-1 in combination with gemcitabine to gemcitabine alone as adjuvant treatment for patients with surgically resected pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed resected ductal pancreatic adenocarcinoma with macroscopic complete resection (R0 and R1). Subjects with neuroendocrine (and mixed type) tumors are excluded.
2. Pancreatic cancer surgical staging: T 1-3, N0-1, M0.
3. Subject should be able to start treatment no later than 12 weeks postsurgery.
4. ≥18 years of age at the time of signing the informed consent form (ICF).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 6. Acceptable hematology parameters:

   * Absolute neutrophil count ≥1500 cell/mm3
   * Platelet count ≥100,000/mm3
   * Hemoglobin (Hgb) ≥9 g/dL 7. Acceptable blood chemistry levels:
   * Aspartate aminotransferase (AST)/ Serum glutamic oxaloacetic transaminase (SGOT) and Alanine transaminase (ALT)/ Serum glutamic -pyruvic transaminase (SGPT) ≤2.5 × upper limit of normal range (ULN)
   * Total bilirubin ≤ Upper Limit of Normal (ULN) (subjects with Gilbert's syndrome can have bilirubin of up to 1.5 x ULN)
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Serum creatinine within upper limits of normal or calculated clearance ≥50 mL/min/1.73 m2. If using creatinine clearance, actual body weight should be used for calculating creatinine clearance (eg, using the Cockroft-Gault formula). For subjects with a Body Mass Index (BMI) >30 kg/m2, lean body weight should be used instead 8. Cancer antigen (CA)19-9 <100 U/mL assessed within 14 days of randomization 9. Acceptable coagulation studies as demonstrated by Prothrombin Time (PT) and Partial Thromboplastin Time (PTT) within normal limits (±15%)

Exclusion Criteria:

1. Prior neo-adjuvant treatment or radiation therapy for pancreatic adenocarcinoma
2. Presence of or history of metastatic pancreatic adenocarcinoma
3. .Any other malignancy within 5 years prior to randomization, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, or nonmelanomatous skin cancer (all treatment of which should have been completed 6 months prior to randomization)
4. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment
5. Known infection with hepatitis B or C, or history of human immunodeficiency virus (HIV) infection, or subject receiving immunosuppressive or myelosuppressive medications that would in the opinion of the investigator, increase the risk of serious neutropenic complications
6. History of allergy or hypersensitivity to nab-paclitaxel or gemcitabine or any of their excipients
7. Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the subject's safety or the study data integrity. These include, but are not limited to:

1).History of connective tissue disorders (eg, lupus, scleroderma, arteritis nodosa) 2).History of interstitial lung disease, slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies 3).History of the following within 6 months prior to Cycle 1 Day 1: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or ECG abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-01; Primary Completion 2021-06 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
DFS | 3 years
  Disease free survival

SECONDARY OUTCOMES:
OS | 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Weijia fang, MD, Principal Investigator — First Affiliated Hospital,Zhejiang University
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China